CLINICAL TRIAL: NCT05840588
Title: Effect of Bifidobacterium Breve PRL2020 (an Amoxicillin-Clavulanate-Resistant Strain) on Gastrointestinal Symptoms and Gut Microbiota Composition in Children Treated With Amoxicillin or Amoxicillin/Clavulanate: Results of a Pediatric, Multicenter, Randomized, Controlled, Prospective Study
Brief Title: Effect of Bifidobacterium Breve PRL2020 (an Amoxicillin-clavulanate-resistant Strain) on Gastrointestinal Symptoms and Gut Microbiota Composition in Children Treated With Amoxicillin or Amoxicillin/Clavulanate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Collaborators: University of Urbino "Carlo Bo" (Other)
Responsible Party: Principal Investigator, Dr. Amjad Khan, Professor, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 77_6settembre2023
Record Dates: First submitted 2023-04-01; First posted 2023-05-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Bifidobacterium breve PRL2020 (Brevicillin®) (Experimental): Patients in this arm will receive Probiotic Bifidobacterium breve PRL2020 (Brevicillin®) (20 billion CFU) 2 sticks/day for 7-10 days (according to antibiotic prescription)in addition to the antibiotic Amoxicillin or Amoxicillin/Clavulanic acid (antibiotic doses: 2-3/day according to physician prescription).
  Interventions: Drug: Antibiotic Treatment; Dietary Supplement: Probiotic Bifidobacterium breve PRL2020 (Brevicillin®) treatment
- Control (Active Comparator): Patients in this arm will receive only antibiotic Amoxicillin or Amoxicillin/Clavulanic acid.
  Interventions: Drug: Antibiotic Treatment

INTERVENTIONS:
Drug: Antibiotic Treatment — Antibiotic Amoxicillin or Amoxicillin/Clavulanic acid
Dietary Supplement: Probiotic Bifidobacterium breve PRL2020 (Brevicillin®) treatment — Probiotic Bifidobacterium breve PRL2020 (Brevicillin®)
  Arms: Probiotic Bifidobacterium breve PRL2020 (Brevicillin®)

SUMMARY:
Amoxicillin or Amoxicillin/Clavulanic acid antibiotic therapy has been shown to be associated with disrupting the microbiota population particularly Bifidobacterium, which may have further GI clinical implications.

The present randomized clinical trial is aimed to assess if probiotic Bifidobacterium breve PRL2020 (Brevicillin®) can help modulate the Bifidobacterium population and its clinical implications after antibiotic Amoxicillin or Amoxicillin/Clavulanic acid antibiotic therapy.

DETAILED DESCRIPTION:
Treatment with Amoxicillin or Amoxicillin/Clavulanic acid is one of the most common antibiotic therapies used against various infections both in children and adults. These antibiotics can create an imbalance in the intestinal microbiota, altering its structure with a reduction in bacterial richness and, more specifically, in the abundance of bifidobacteria. This opened the window for further evaluations of the effect of this antibiotic combination on the composition of gut microbiota. The alteration can lead to intestinal symptoms such as pain, bloating, abdominal distension, flatulence, diarrhea, and constipation. In study by L. Mancabelli et al. (2021), Bifidobacterium breve PRL2020 has shown greatest resistance to Amoxicillin and Amoxicillin/Clavulanic acid. Currently available scientific data, however, have not yet analyzed the ability of B. breve PRL2020 to counteract the reduction of bifidobacteria that may occur in the human gut during the antibiotic therapy with Amoxicillin or Amoxicillin/Clavulanic acid, and neither its ability to avoid the consequent clinical relapse.

The purpose of this randomized, controlled (untreated group), prospective, multicentre, single-center, non-profit study will be to evaluate the efficacy and safety of the administration of Bifidobacterium breve PRL2020 (Brevicillin®) in pediatric patients (> 3 -12 years of age), treated with the antibiotic Amoxicillin or Amoxicillin/Clavulanic acid, in the improvement of the symptoms due to the pharmacological treatment and in the contrast of the fall of the Bifidobacterium cluster.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3-12 years, of either gender, with a bacterial infection and the use of antibiotic therapy with Amoxicillin or Amoxicillin/clavulanic acid under a Physician's prescription.

Exclusion Criteria:

* Presence of neurological, oncological (also past), malformative, and/or autoimmune pathology
* Suspected or presumed allergy to the substance contained in the probiotic formula
* Using any type of probiotic product in the three months before the enrollment or during the trial
* Lack of parental consent to participate in the study

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Incidence of antibiotic-associated diarrhea (AAD) | 7-10 days (according to antibiotic prescription)
  Assessment of diarrhea occurring during antibiotic treatment with amoxicillin or amoxicillin/clavulanic acid.
  AAD will be counted starting from a single episode of diarrhea and not only after three or more episodes in one day, differing from the standard AAD definition.
Incidence of gastrointestinal symptoms other than diarrhea | 7-10 days (according to antibiotic prescription)
  Evaluation of gastrointestinal symptoms related to antibiotic therapy, including constipation, nausea, vomiting, abdominal cramps, bloating, and loss of appetite. These will be recorded daily by parents or legal guardians during the antibiotic course.

SECONDARY OUTCOMES:
Change in gut microbiota diversity following probiotic and antibiotic treatment | 7-10 days (according to antibiotic prescription)
  Change in gut microbiota composition and diversity assessed by 16S rRNA sequencing of stool samples collected during and after the treatment period. Alpha diversity (Shannon index) and relative abundance of Bifidobacterium genus will be calculated and compared between groups.
Tolerability of probiotic treatment | 7-10 days (according to antibiotic prescription)
  Number of participants rated as having "good" or "excellent" tolerability to probiotic treatment, as assessed by the physician at the end of antibiotic therapy. Tolerability will be evaluated based on clinical observation and parental report of side effects (e.g., nausea, abdominal discomfort, rash).
Adherence to probiotic treatment | 7-10 days (according to antibiotic prescription)
  Percentage of participants who completed ≥80% of the prescribed probiotic doses during the antibiotic treatment period, as assessed by returned product count and parental report.

CONTACTS AND LOCATIONS:
Locations (1):
- Università di Urbino Carlo Bo, Urbino, PU (Pesaro E Urbino), Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mancabelli L, Mancino W, Lugli GA, Argentini C, Longhi G, Milani C, Viappiani A, Anzalone R, Bernasconi S, van Sinderen D, Ventura M, Turroni F. Amoxicillin-Clavulanic Acid Resistance in the Genus Bifidobacterium. Appl Environ Microbiol. 2021 Mar 11;87(7):e03137-20. doi: 10.1128/AEM.03137-20. Print 2021 Mar 11. PMID 33483308
- [Background] Bartlett JG. Clinical practice. Antibiotic-associated diarrhea. N Engl J Med. 2002 Jan 31;346(5):334-9. doi: 10.1056/NEJMcp011603. No abstract available. PMID 11821511
- [Background] Salvo F, Polimeni G, Moretti U, Conforti A, Leone R, Leoni O, Motola D, Dusi G, Caputi AP. Adverse drug reactions related to amoxicillin alone and in association with clavulanic acid: data from spontaneous reporting in Italy. J Antimicrob Chemother. 2007 Jul;60(1):121-6. doi: 10.1093/jac/dkm111. Epub 2007 Apr 21. PMID 17449881
- [Background] Caron F, Ducrotte P, Lerebours E, Colin R, Humbert G, Denis P. Effects of amoxicillin-clavulanate combination on the motility of the small intestine in human beings. Antimicrob Agents Chemother. 1991 Jun;35(6):1085-8. doi: 10.1128/AAC.35.6.1085. PMID 1929247
- [Background] Yang L, Bajinka O, Jarju PO, Tan Y, Taal AM, Ozdemir G. The varying effects of antibiotics on gut microbiota. AMB Express. 2021 Aug 16;11(1):116. doi: 10.1186/s13568-021-01274-w. PMID 34398323
- [Background] Liu L, Wang Q, Lin H, Das R, Wang S, Qi H, Yang J, Xue Y, Mao D, Luo Y. Amoxicillin Increased Functional Pathway Genes and Beta-Lactam Resistance Genes by Pathogens Bloomed in Intestinal Microbiota Using a Simulator of the Human Intestinal Microbial Ecosystem. Front Microbiol. 2020 Jun 4;11:1213. doi: 10.3389/fmicb.2020.01213. eCollection 2020. PMID 32582117
- [Background] Duranti S, Lugli GA, Milani C, James K, Mancabelli L, Turroni F, Alessandri G, Mangifesta M, Mancino W, Ossiprandi MC, Iori A, Rota C, Gargano G, Bernasconi S, Di Pierro F, van Sinderen D, Ventura M. Bifidobacterium bifidum and the infant gut microbiota: an intriguing case of microbe-host co-evolution. Environ Microbiol. 2019 Oct;21(10):3683-3695. doi: 10.1111/1462-2920.14705. Epub 2019 Jun 20. PMID 31172651